CLINICAL TRIAL: NCT01773434
Title: A Phase 1 Study of MORAb-004 in Patients With Solid Tumor
Brief Title: A Phase 1 Study of MORAb-004 in Patients With Solid Tumor (Study: MORAb-004-J081-103)
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Eisai Co., Ltd. (Industry)
Responsible Party: Sponsor
Organization: Eisai Inc. (Industry)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: MORAb-004-J081-103
Record Dates: First submitted 2013-01-17; First posted 2013-01-23 (Estimated); Last update posted 2016-11-10 (Estimated); Status verified 2016-11

CONDITIONS: Solid Tumor
MeSH Terms: interventions — ontuxizumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- MORAb-004 (Experimental)
  Interventions: Drug: MORAb-004

INTERVENTIONS:
Drug: MORAb-004 — MORAb-004 5 mg/mL is administered as an intravenous infusion (IV) in an escalating dose design and will not be escalated or de-escalated in individual participants.
  Part 1 (Dose escalation): 4 weekly administrations of 2, 4, 8, and 12 mg/kg in four different cohorts on Days 1, 8, 15, and 22 of a 4-week cycle (28 days).
  Part 2 (Cohort expansion): 4 and 8 mg/kg on Days 1, 8, 15, and 22 of a 4-week cycle (28 days) and 12 mg/kg biweekly administration on Days 1 and 15 of a 4-week cycle in different cohorts. The dosages in Part 2 can be amended considering the results of Part 1.

SUMMARY:
This is a multicenter, multiple doses, open-label Phase 1 study of MORAb-004 in subjects with solid tumors. Subjects may have any solid tumor without intracranial involvement or metastases that has failed standard chemotherapy.

This study will be conducted in 2 parts: 1) Part 1 will be the dose escalation portion of this study to assess the tolerability and the safety profile of MORAb-004. Dose will escalate in different cohorts as follows: 2, 4, 8 and 12 mg/kg weekly dosing each as a 4-week cycle with no intra-subject escalation. Individual participants may have additional cycles at the same dose until disease progression unless the participants meet the discontinuation criteria.

2) Part 2 will comprise cohort expansions to further characterize the safety and tolerability of MORAb-004 and to assess preliminary efficacy and the pharmacokinetic/pharmacodynamic relationship of MORAb-004 in gastric cancer and hepatocellular carcinoma (HCC). Three dose levels will be expanded based on the safety profile that was obtained in the dose escalation portion of this study (Part 1): 4 mg/kg (administered on a weekly basis), 8 mg/kg (administered on a weekly basis) and 12 mg/kg (administered every OTHER week).

ELIGIBILITY:
Inclusion criteria:

1. Provide written informed consent,
2. Japanese male and female subjects aged at 20 or older at informed consent,
3. Have malignant solid tumor, without intracranial involvement or metastasis, diagnosed by standard pathology criteria that has failed or are resistant to standard chemotherapy,
4. Performance status (PS) is 0 to 1 by Eastern Cooperative Oncology Group,
5. With no carry-over effect and no adverse drug reaction of prior treatment which may affect the safety evaluation of MORAb-004, except for Grade 1 or 2 neuropathy and alopecia,
6. Survival expectation is 12 weeks or longer after starting MORAb-004 administration

Exclusion criteria:

1. Have clinically significant cardiovascular disease,
2. Scheduled for laparotomic surgery due to trauma or other reasons for during the study,
3. Have clinically significant hemorrhagic event or history, or event with high risk of hemorrhage,
4. Receiving chronic systemic anticoagulation,
5. Have evidence of other active invasive malignancy
6. Females who are lactating or pregnant at Screening or Baseline

Min Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 46 (Actual)
Dates: Start 2012-12; Primary Completion 2016-07 (Actual); Study Completion 2016-10 (Actual)

PRIMARY OUTCOMES:
Tolerability and Safety | Up to 30 months
  Tolerability and the safety profile of multiple intravenous (IV) infusions of MORAb-004 in Japanese participants with solid tumors.

SECONDARY OUTCOMES:
Maximum Tolerated Dose (MTD)- Part I | Up to 30 months
  Maximum tolerated dose (MTD) as defined by dose limiting toxicities (DLTs) within the administered range.
Optimal Biologic Dose (OBD)- Part II | Up to 30 months

CONTACTS AND LOCATIONS:
Overall Officials: Ryo Nakajima, Study Director — Eisai Co., Ltd.
Locations (4):
- Japan (4):
  - Chikusa-ku, Aichi-ken
  - Kashiwa, Chiba
  - Nagaizumi-cho, Shizuoka
  - Chuo-ku, Tokyo

REFERENCES:
- [Derived] Doi T, Aramaki T, Yasui H, Muro K, Ikeda M, Okusaka T, Inaba Y, Nakai K, Ikezawa H, Nakajima R. A phase I study of ontuxizumab, a humanized monoclonal antibody targeting endosialin, in Japanese patients with solid tumors. Invest New Drugs. 2019 Oct;37(5):1061-1074. doi: 10.1007/s10637-018-0713-7. Epub 2019 Jan 9. PMID 30623276